CLINICAL TRIAL: NCT02824614
Title: Effect of the Natural Sweeteners Erythritol and Xylitol on Gut Microbiota and Glucose Metabolism in Obese Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Poly Gut
Record Dates: First submitted 2016-06-27; First posted 2016-07-06 (Estimated); Last update posted 2025-07-20 (Actual); Status verified 2020-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Xylitol; Erythritol

STUDY DESIGN:
Intervention Model Description: Mullti-center trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): 20 obese, non-diabetic candidates will serve as control-group. All assessments are carried out just as in the intervention groups.
- E967-Xylitol (Active Comparator): 20 obese, non-diabetic candidates will receive a daily dose of 24g of xylitol.
  Interventions: Dietary Supplement: E967-Xylitol
- E968-Erythritol (Active Comparator): 20 obese, non-diabetic candidates will receive a daily dose of 36g of erythritol.
  Interventions: Dietary Supplement: E968-Erythritol

INTERVENTIONS:
Dietary Supplement: E967-Xylitol
  Other Names: Xylitol
  Arms: E967-Xylitol
Dietary Supplement: E968-Erythritol
  Other Names: Erythritol
  Arms: E968-Erythritol

SUMMARY:
Sugar alcohols such as xylitol and erythritol are increasingly popular as sugar substitutes in the food industry and are also recommended to diabetic patients. Both substances are already in use in the food industry and are freely available. Since the 1970s, beneficial effects on oral health could be demonstrated as oral bacteria were influenced positively. Animal studies showed an increase in gut Clostridium perfringens after xylitol intake; certainly a non-desirable effect. However, studies on effects of erythritol and xylitol on the human gut microbiota are lacking so far. In this trial, investigators aim to examine whether gut microbiota and glucose tolerance can be influenced by polyol intake in a non-diabetic but obese cohort.

ELIGIBILITY:
Inclusion Criteria:

* Obese volunteers (BMI > 30kg/m2)
* Aged 18- max. 55 years
* Otherwise healthy.

Exclusion Criteria:

* Known cardiovascular disease
* Diabetes mellitus
* Arterial Hypertension with medication
* Dyslipidaemia with medication
* Known chronic hepatic disease (NASH, hepatitis).
* Known renal disease: kidney failure
* Pregnancy
* Intake of proton pump inhibitors (PPIs) on a regular basis
* Intake of antibiotics within the last 3 months before inclusion
* Intake of pro or prebiotics
* Chronical diseases of the gastrointestinal tract, history of gastrointestinal surgery with major changes to the gastrointestinal tract
* Substance abuse, alcohol abuse.
* Inability to follow procedures due to psychological disorders, dementia or insufficient knowledge of project language (German).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance measured with oral glucose tolerance test | change from baseline to 8 weeks after polyol intake

SECONDARY OUTCOMES:
Human gut microbiota composition measured with metagenomic shotgun sequencing | change from baseline to 8 weeks after polyol intake
Gut microbial-related metabolites in feces | change from baseline to 8 weeks after polyol intake
  Metabolomic analysis of the bacterial metabolites present in the feces by combining nuclear magnetic resonance (1H-NMR) and mass spectrometry
Gastrointestinal tolerance assessed by questionnaire | change from baseline to 8 weeks after polyol intake
  Gastrointestinal Symptoms Rating Scale (Svedlund et al)
Gut microbial-related metabolites in urine | change from baseline to 8 weeks after polyol intake
  Metabolomic analysis of the bacterial metabolites present in the urine by combining nuclear magnetic resonance (1H-NMR) and mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, MD, Study Chair — St. Claraspital klinische Forschungsabteilung
Locations (3):
- Department of Endocrinology, Morbid Obesity and Preventive Medicine, Oslo University Hospital, Oslo, Norway
- Endoscopic and Minimally Invasive Surgery Clinic of Stavropol State Medical University, Stavropol, Russia
- St Claraspital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided